CLINICAL TRIAL: NCT02021266
Title: Single Patient Expanded Access Protocol: Phase I/II Pilot Study of Mixed Chimerism to Treat Inherited Metabolic Disorders
Brief Title: Single Patient Expanded Access Protocol: Metabolic Boost
Acronym: Boost
Status: No longer available | Type: Expanded Access
Sponsor: Talaris Therapeutics Inc. (Industry)
Collaborators: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: ICT-14070-120611-Exp Access
Record Dates: First submitted 2013-12-19; First posted 2013-12-27 (Estimated); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Metachromatic Leukodystrophy
MeSH Terms: conditions — Leukodystrophy, Metachromatic

INTERVENTIONS:
Biological: Enriched Hematopoetic Stem Cell Infusion — Enriched Hematopoetic Stem Cell Infusion

SUMMARY:
This is a single patient expanded access protocol to investigate the effects of a second dose of facilitating cell-enhanced hematopoietic stem cell product.

DETAILED DESCRIPTION:
Hematopoietic stem cell transplantation (HSCT) has been established as an important therapeutic option for patients with a variety of inherited metabolic disorders (IMD). The potential life-threatening complications of conventional myeloablative HSCT have limited its application. Additionally, conventional HSCT is only available to the small minority of medically suitable candidates who have histocompatibility leukocyte antigen (HLA)-identical siblings to donate bone marrow or mobilized peripheral blood stem cells.

Donor mobilized peripheral blood stem cells or bone marrow will be processed via a novel technology to deplete mature immune cells while retaining hematopoietic stem cells (HSC) and graft facilitating cells (FC).

A now-standard reduced intensity, nonmyeloablative recipient conditioning regimen will be used to promote mixed allogeneic chimerism, thereby significantly reducing morbidity and mortality.

These two enhancements are intended to significantly improve the benefit:risk ratio of HSCT for patients with IMDs. If successful, transplantation will become a more feasible option for patients without HLA-identical siblings to donate stem cells, and could be offered to patients early in disease progression.

The objective for the study is to establish chimerism following reduced intensity conditioning with no grade III/IV graft-versus-host disease (GVHD). The primary endpoint we will follow is production of the missing enzyme at ≥ 10% of the normal level at day 180 post-transplant as for investigational new drug (IND) 14070. This expanded access protocol details the approach to providing a second dose of the product.

ELIGIBILITY:
Inclusion Criteria:

Subject was previously enrolled and qualified for transplant under IND 14070. Subject must be free from infection and have normal liver, kidney, heart and pulmonary function to proceed to a second transplant.

1. Patient must have adequate function of other organ systems as measured by:

   * Creatinine < 2.0 mg/dl and creatinine clearance ≥60 cc/min/1.73m2. Newborns must have a creatinine clearance > 25 cc/min. For babies < 3 months of age, the raw value on GFR must be > 1 cc/kg/min.
   * Hepatic transaminases (ALT/AST) 2.5 x normal, bilirubin <2.0mg/dl
   * Normal cardiac function by echocardiogram or radionuclide scan (ejection fraction or shortening fraction >80% of normal value for age)
   * Pulmonary function tests (PFT) demonstrating forced expiratory volume at one second (FEV1) of >50% of predicted for age. If child is too young or unable to perform PFTs, crying vital capacity result of >50% of normal value for age or resting pulse oximeter >92% on room air or clearance by pulmonologist will be required.
2. Patient, and parent, or legal guardian must have given written informed consent according to FDA guidelines.
3. Patient must have a minimum life expectancy of at least 6 months.
4. Female patients of childbearing potential cannot be pregnant or lactating/breast-feeding and must be either surgically sterile, postmenopausal (no menses for the previous 12 months), or must be practicing an effective method of birth control as determined by the investigator (e.g., oral contraceptives, double barrier methods, hormonal injectable or implanted contraceptives, tubal ligation, or partner with vasectomy).
5. Recipient screening to include glomerular filtration rate (GFR), chest X-ray (CXR), hepatic and renal chemistries, coagulation studies, pulmonary function testing, and ECHO if clinically relevant, chimerism testing, type and screen, and enzyme levels within 30 days of retransplant.

Exclusion Criteria:

1. Uncontrolled seizures, apnea, evidence of recurrent or uncontrolled aspiration, or need for chronic mechanical ventilation.
2. Subject must not have had previous radiation therapy that would preclude total body irradiation (TBI) (as determined by radiation therapist)
3. Uncontrolled infection or severe concomitant diseases, which in the judgment of the Principal Investigator, could not tolerate reduced intensity transplantation.
4. Subject with a positive human immunodeficiency virus (HIV) antibody test result
5. Subject who are pregnant, as indicated by a positive serum human chorionic gonadotropin (HCG) test
6. Subject whose only donor is pregnant at the time of intended transplant
7. Subject of childbearing potential who are not practicing adequate contraception as defined by the investigator at the site
8. Jehovah's witnesses being unwilling to be transfused
9. Patient that have any comorbid condition which, in the view of the Principal Investigators, renders the patient at too high a risk from treatment complications and regimen related morbidity/mortality.
10. Insufficient funds for bone marrow processing.

Sex: Female
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne T Ildstad, MD, Study Director — Talaris Therapeutics Inc.
Locations (1):
- Duke University, Durham, North Carolina, United States